CLINICAL TRIAL: NCT04150627
Title: Effect of Breathing Maneuvers on Peripheral Glucose Metabolism
Acronym: RESPI01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 039/2019B02
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2019-10

CONDITIONS: Vagus Nerve Stimulation; Insulin Sensitivity; Deep Breathing Maneuver
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deep breathing (Active Comparator)
  Interventions: Other: deep breathing
- normal breathing (No Intervention)

INTERVENTIONS:
Other: deep breathing — Deep breathing maneuver to increase parasympathetic nerve activity
  Arms: deep breathing

SUMMARY:
Two important mechanisms play a major role in the pathogenesis of type 2 diabetes: insulin resistance of the target tissues and the impaired insulin secretion from pancreatic β-cells. Postprandial factors (such as insulin) are perceived by the human brain and induce signals that regulate glucose metabolism via the parasympathetic nervous system.

Deep breathing exercise can increase parasympathetic nerve activity. Heart rate variability (HRV) in healthy people can be significantly increased by deep breathing maneuvers, indicating a shift from sympathetic activity to parasympathetic activity.

The hypothesis is that this postprandial shift results in a change in peripheral glucose metabolism. In turn, the increased parasympathetic activity could potentially result in a change in postprandial insulin sensitivity or secretion.

To test this hypothesis, this study investigates the effect of deep breathing exercise versus normal breathing on insulin sensitivity, on insulin secretion, glucose tolerance, resting energy expenditure, and on parasympathetic tone (analysis of heart rate variability).

ELIGIBILITY:
Inclusion Criteria:

* HbA1c <6.5%
* Must be able to understand the explanations of the study and the instructions

Exclusion Criteria:

* Any relevant (according to investigator's judgment) cardiovascular disease
* Neurological and psychiatric disorders
* Diabetes mellitus
* Asthma

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Whole body insulin sensitivity | 0-120 min
  Insulin sensitivity will be assessed by a 75g OGTT

SECONDARY OUTCOMES:
Insulin secretion | 0-120 min
  Insulin secretion will be assessed by a 75g OGTT
Glucose tolerance | 0-120 min
  Glucose tolerance will be assessed by a 75g OGTT
Resting energy expenditure | 140-160 min after start of breathing maneuver
  Resting energy expenditure will be assessed by indirect calorimetry
Heart rate variability | -35 - 120 min
  Heart rate variability will be assessed from continuous ecg recordings

CONTACTS AND LOCATIONS:
Overall Officials: Martin Heni, MD, Principal Investigator — University Hospital Tübingen
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No